CLINICAL TRIAL: NCT07298486
Title: Impact of Robotic Glove Use on Quality of Life, Grip Strength and Fine Motor Control in ALS: A Pilot Study
Brief Title: Impact of Robotic Glove Use on Quality of Life, Grip Strength and Fine Motor Control in ALS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Kayla Chomko, Rehabilitation Director, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-320-NSU; 337263 (Other Grant/Funding Number: Husman Study Fund)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; ALS; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic Glove Intervention (Experimental): Participants with initiate robotic glove use 5 days / week , 1x/day for 20 minutes
  Interventions: Device: Robotic Glove Use

INTERVENTIONS:
Device: Robotic Glove Use — The participant or caregiver will don the robotic glove and power on the device. A timer will be set for 20 minutes. The participant will sit comfortably at a table with their elbow supported on the table. When the time is complete, the robotic glove will be powered off and the glove removed. The PI and/or study team will be present throughout the first 2 sessions and 2 sessions midway into the 8 week study period to monitor for discomfort, fatigue or any additional patient reported symptoms. The participant will complete a total of 40 intervention sessions.
  Weekly telephone calls will be conducted by study team members to ensure compliance with the protocol, the robotic glove is working properly and answer any questions the participant or caregiver may have.

SUMMARY:
The goal of this clinical trial is to determine the impact of robotic glove use on quality of life, grip strength and fine motor control in participants with Amyotrophic Lateral Sclerosis (ALS). This will provide valuable insights into how an assistive technology intervention can influence functional ability in daily tasks and enhance overall well-being in individuals impacted by ALS.

Participants will attend 3 in-person clinic visits (BASE, 4 week and 8 week visit) and 2 Telehealth visits (occurring 24 hours after BASE and 4 week visit). The in-person clinic visits will include assessments by either a physical or occupational therapist, followed by assessments and scoring of grip strength, various fine motor strength assessments of affected hand, fine motor coordination assessment of the affected hand and various quality of life scales.

The participant will be fitted and measured for the appropriately sized robotic glove. Once the fit is confirmed, both the participant and caregiver will receive education on how to don and doff the glove, power it on and off, and follow the study protocol. Once they demonstrate understanding and independence with these steps, the intervention will begin.

The robotic glove intervention consists of either the participant or caregiver donning the glove and powering it on. A timer will be set for 20 minutes. The participant will sit comfortably at a table with their elbow supported on the table. The PI and/or member of the study team will be present throughout the 20 minute session to monitor for discomfort, fatigue or any additional patient reported symptoms. Once the time is complete, the robotic glove will be powered off and the glove removed. The participant and caregiver will be instructed to perform this one time daily, for 5 days per week for a total of 8 weeks. The PI and study team members will be available for any questions via iPhone or e-mail throughout this time period.

The Telehealth visits will consist of synchronous video and audio via the Zoom application. The PI and/or study team members will monitor the set up, application and powering on of the Robotic Glove. The treatment of 20 minutes will be monitored and any questions the participant or caregiver have will be answered. This visit's goal is to ensure compliance and proper application of the robotic glove.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the impact of robotic glove use on quality of life, grip strength and fine motor control in participants with ALS. The study population includes 5 participants with a diagnosis of ALS, aged 18-99.

Once consent and enrollment is complete, the participant will be measured for their robotic glove size on day of enrollment. The robotic glove is a rehabilitation device that fits over the participants fingers and is secured through velcro straps. It delivers passive range of motion through an air pump that facilitates finger flexion and extension.

Measurements will be performed with a standard tape measure. The following 3 measurements will be taken of the participants affected hand:

1. Hand width: determined by the base of the 1st metacarpal to distal end of 5th metacarpal
2. Hand length: determined by lunate to distal end of distal phalanx of digit 3
3. Middle finger circumference: determined by the circumference of the distal end of proximal phalanx of digit

The proper size robotic glove will be obtained and the BASE clinic visit will be scheduled.

Each participant will then attend three (3) in=person clinic visits and participate in two (2) telehealth visits. The clinic visits will take place at three time points: baseline (BASE), 4 weeks after the start date (4W), and post-intervention at 8 weeks (POST). The BASE visit is expected to last 60 minutes. The 4W and POST visits are expected to last 30 minutes.

Outcome measures that will be assessed at each in person clinic visit include:

1. Amyotrophic Lateral Sclerosis Quality of Lift Short Form (ALS QOL short form)
2. EuroQOL-5D (EQ-5D)
3. Grip Strength
4. 9 Hole PEG test
5. Tip-to-Tip pinch strength
6. Palmar pinch strength
7. Key pinch strength
8. Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) and its Gross motor and fine motor sub-scales (GMS) (FMS)

BASE visit:

The Base visit will consist of above mentioned assessments followed by training of both patient and caregiver on how to don and doff the robotic glove. The PI and/or study team will complete the training, followed by monitoring the patient and caregiver successfully applying the Robotic glove. The PI will manually set the robotic glove for passive mode with a 6 second on time and 6 second off time. Once the participant and caregiver are able to successfully demonstrate application and removal of the robotic glove, including powering on and off the robotic glove, the robotic glove intervention will commence.

ROBOTIC GLOVE INTERVENTION: The participant or caregiver will don the robotic glove and power on the device. A timer will be set for 20 minutes. The participant will sit comfortably at a table with their elbow supported on the table. The PI and/or study team member will be present throughout the 20 minute session to monitor for discomfort, fatigue or any additional patient reported symptoms. Once the time is complete, the robotic glove will be powered off and the glove removed.

The participant and caregiver will be instructed to perform this one time daily, for 5 days per week for a total of 8 weeks. The PI and Co-PI will be available for any questions via iPhone or e-mail throughout this time period.

Telehealth Visit #1 (TH1):

This visit will commence on day 2 and will take approximately 30 minutes. A telehealth appointment will be set up with the participant and their caregiver 24 hours after the baseline visit. This will consist of synchronous video and audio via the Zoom application. The PI and/or Co-PI will monitor the set up, application and powering on of the Robotic Glove. The treatment of 20 minutes will be monitored and any questions the participant or caregiver have will be answered. This visit's goal is to ensure compliance and proper application of the robotic glove.

4W visit: The 4W visit will consist of above mentioned assessments (#1-8) as previously described in the BASE visit and will be completed in person. This is expected to last 30 minutes

Telehealth Visit #2 (TH2):

This visit will commence 24 hours after visit 4W and will mimic TH1.

POST visit:

This will occur during week 8 once all 40 intervention sessions have been completed. The participant and caregiver will be brought in to the clinic and assessments 1-8 will be completed.

This will conclude the study intervention.

Weekly telephone calls will be conducted by study personnel to ensure compliance with the protocol, the robotic glove is working properly and answer any questions the participant or caregiver may have.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically possible, probable or definite amyotrophic lateral sclerosis by the treating neurologist
* Have a caregiver that is willing and present to assist with application of robotic glove
* Reports fine motor deficits or grip strength deficits in at least 1 hand
* Demonstrates > or = 3 lbs. of Grip strength as measured by a dynamometer on affected hand AND/OR Demonstrates Fine motor deficits and has > or = 1 lb. of pinch strength (tip to tip, three jaw chuck, or lateral key pinch) as measured by pinch gauge dynamometer
* Demonstrates a loss of at least 3 lbs. of Grip strength OR 1lb. of pinch strength over a minimum of 1 month period in affected hand
* Stable dose of efficacious medications for 30 days.

Exclusion Criteria:

* History of Rheumatoid Arthritis
* History of Depuytren's contracture
* Open wound at affected hand where robotic glove will be placed
* History of Trigger Finger
* Complete loss of sensation at the affected hand where robotic glove will be placed
* History of Carpal Tunnel Syndrome
* Prior or current use of robotic glove
* Active physical or occupational therapy treatment interventions on affected hand

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
ALS-Specific Quality of Life Questionnaire - Short Form | Baseline, 4 weeks, 8 weeks
  is a validated, disease-specific questionnaire designed to assess quality of life in individuals with ALS. It provides a concise measure of key domains such as emotional well-being, physical symptoms, social interaction, and existential concerns. The short-form version reduces patient burden while maintaining strong reliability and sensitivity to changes in health status over time.

SECONDARY OUTCOMES:
EuroQOL-5D | Baseline, 4 weeks and 8 weeks
  a standardized, patient-reported outcome measure used to assess health-related quality of life. It evaluates five key dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each rated by level of severity. It also includes a visual analog scale (VAS) where patients rate their overall health from 0 to 100.
Grip Strength | Baseline, 4 weeks, 8 weeks
  Grip strength is measured in pounds utilizing a handheld dynamometer. The participant will be asked to perform maximum grip strength by squeezing a handheld dynamometer over 3 seconds, 3 reps and the average will be taken.
Finger tip to tip pinch strength | baseline, 4 weeks, 8 weeks
  Fingertip-to-tip pinch strength is measured by having the patient press the tip of their thumb and the tip of their index finger together against a pinch gauge. The patient applies maximal pressure, and the device records the force generated. The participant will be asked to complete this 3 times and the average will be taken.
Palmar pinch strength | Baseline, 4 weeks and 8 weeks
  Palmar pinch strength (also called three-jaw chuck pinch) measures the force generated when the thumb presses against the pads of the index and middle fingers. Using a pinch gauge, the participant is asked to squeeze as firmly as possible. Three trials are performed, and the average is recorded. This measure reflects the ability to perform everyday tasks requiring precision and control, such as holding a key, buttoning clothes, or picking up small objects.
Key Pinch Strength | Baseline, 4 weeks and 8 weeks
  This test reflects functional hand strength used in tasks like turning a key, gripping a card, or opening a door. Using a pinch gauge, the participant is asked to place the gauge between the thumb pad and side of the index finger and pinch as hard as possible. 3 trials are performed and the average force is recorded.
9 Hole PEG test | Baseline, 4 weeks and 8 weeks
  A standardized assessment of finger dexterity and fine motor coordination. The participant is asked to place nine pegs into nine holes and then remove them as quickly as possible, using their affected hand. The time taken to complete the task is recorded. Faster times indicated improved manual dexterity.
Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) | Baseline, 4 weeks and 8 weeks
  It evaluates 12 items across four domains: bulbar (speech, swallowing), fine motor (handwriting, dressing), gross motor (walking, climbing stairs), and respiratory function (breathing, dyspnea).
  Each item is scored from 0 (worst) to 4 (normal), giving a total score from 0 to 48, with higher scores indicating better function. It's used to track disease progression and assess response to treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Kayla Chomko, PT, DPT, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, David and Cathy Husman Neuroscience Institute, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All 5 participants baseline assessments, 4 week assessments and post assessments will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD will be available 12 months after publication of the primary results and for a period of 5 years.
Access Criteria: De-identified IPD will be shared with qualified researchers upon reasonable request, subject to review by the study investigators and execution of a data use agreement.

REFERENCES:
- [Background] Felgoise SH, Feinberg R, Stephens HE, Barkhaus P, Boylan K, Caress J, Clawson LL, Elman L, Goutman SA, Mccluskey L, Russell J, Tiryaki E, Weiss M, Simmons Z. Amyotrophic lateral sclerosis-specific quality of life-short form (ALSSQOL-SF): A brief, reliable, and valid version of the ALSSQOL-R. Muscle Nerve. 2018 Nov;58(5):646-654. doi: 10.1002/mus.26203. Epub 2018 Oct 19. PMID 30028537
- [Background] Hayden CD, Murphy BP, Hardiman O, Murray D. Measurement of upper limb function in ALS: a structured review of current methods and future directions. J Neurol. 2022 Aug;269(8):4089-4101. doi: 10.1007/s00415-022-11179-8. Epub 2022 May 25. PMID 35612658
- [Background] Wang T, Liu Z, Gu J, Tan J, Hu T. Effectiveness of soft robotic glove versus repetitive transcranial magnetic stimulation in post-stroke patients with severe upper limb dysfunction: A randomised controlled trial. Front Neurol. 2023 Jan 11;13:887205. doi: 10.3389/fneur.2022.887205. eCollection 2022. PMID 36712422
- [Background] Yamakawa I, Yamada A, Sonoda Y, Wakita K, Nishioka T, Harada Y, Ogawa N, Kitamura A, Sanada M, Tani T, Imai S, Urushitani M. Occupational therapy using a robotic-assisted glove ameliorates finger dexterity and modulates functional connectivity in amyotrophic lateral sclerosis. J Clin Neurosci. 2023 Jan;107:144-149. doi: 10.1016/j.jocn.2022.11.004. Epub 2022 Nov 18. PMID 36411175